CLINICAL TRIAL: NCT05712083
Title: Clinical Trial for the Safety and Efficacy of BCMA CAR-T Cell Therapy for Newly Diagnosed Multiple Myeloma
Brief Title: A Study of BCMA CAR-T Cell Therapy for Newly Diagnosed Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210024C-R4
Record Dates: First submitted 2023-01-31; First posted 2023-02-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma; New Diagnosis Tumor
Keywords: BCMA CAR-T; Multiple Myeloma; New Diagnosis
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This is a single arm clinical trial.
  Interventions: Drug: BCMA CAR-T cells

INTERVENTIONS:
Drug: BCMA CAR-T cells — Each subject receive BCMA CAR T-cells by intravenous infusion
  Other Names: BCMA CAR-T cells injection

SUMMARY:
Clinical Trial for the Safety and Efficacy of BCMA CAR-T Cell Therapy for Newly Diagnosed Multiple Myeloma

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for newly diagnosed multiple myeloma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 40 patients will be enrolled. Primary objective is to explore the safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* 1.Age and gender unlimited;
* 2.According to the IMWG2014 standard, diagnosis as multiple myeloma;
* 3.According to the MSMART 3.0 standard, it is defined as a high-risk multiple myeloma;
* 4.Abnormal plasmocyte BCMA expression positive;
* 5.Echocardiography shows the left ventricular ejection score (LVEF) ≥50%;
* 6.The subject has no lung activity infection;
* 7.Expected life time is more than 3 months;
* 8.ECOG score 0-2 score;
* 9.Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* 1.Patients with the history of epilepsy or other CNS disease;
* 2.Patients with prolonged QT interval time or severe heart disease;
* 3.Pregnant or breastfeeding;
* 4.Active infection with no cure;
* 5.Patients with active hepatitis B or C infection;
* 6.Previously treated with any genetic therapy;
* 7.The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8.Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
* 9.Those who suffer from other uncontrolled diseases are not suitable to join the study;
* 10.HIV infection;
* 11.Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after BCMA CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Baseline up to 2 years after BCMA CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Multiple Myeloma (MM), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = sCR+CR+VGPR+PR+MR) at Month 6, 12, 18 and 24
Complete response rate(CRR) | Baseline up to 2 years after BCMA CAR T-cells infusion
  Proportion of subjects who achieved morphological complete response (CR) and complete response with hematologic incomplete recovery (CRi)
Partial response Rate (PRR) | Up to 2 years after BCMA CAR T-cells infusion
  Proportion of subjects who achieved a partial response (PR)
Overall survival | Up to 2 years after BCMA CAR T-cells infusion
  Death from any cause from the beginning of cell transfusion

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China